CLINICAL TRIAL: NCT02263196
Title: Mashhad University of Medical Sciences
Brief Title: The Efficacy of Alcohol After Betadine and Combination of Alcohol and Betadine on Inflammation Vascular Access
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, rajabpoor, Mashhad University of Medical Sciences, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 921839
Record Dates: First submitted 2014-09-26; First posted 2014-10-13 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Complication of Hemodialysis
MeSH Terms: interventions — Ethanol; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alcohol and povidone iodine (Experimental): the efficacy of combination of alcohol and povidone iodine on inflammation related to vascular access
  Interventions: Other: Alcohol and povidone iodine
- combination of alcohol and betadin (Experimental): the efficacy of combination of alcohol and povidone iodine on infection related to vascular access
  Interventions: Other: combination of alcohol and betadin

INTERVENTIONS:
Other: Alcohol and povidone iodine — using from Alcohol and povidone iodine for prevention of inflammation
  Arms: alcohol and povidone iodine
Other: combination of alcohol and betadin — using from combination Alcohol and povidone iodine for prevention of inflammation
  Arms: combination of alcohol and betadin

SUMMARY:
The purpose of this study was to compare the efficacy of combination of alcohol and povidone iodine 10% and Alcohol 70% after povidone iodine 10% on inflammation and infection related to vascular access area in hemodialysis patients.

DETAILED DESCRIPTION:
These cases were identified from patient that lack of specific diseases; Non-use of antibiotics or immunosuppressive drugs. That the participants will be selected using convenience sampling method and randomly divided into three groups: combination of alcohol and povidone iodine 10%, Alcohol after and control groups. In the Intervention in one group the vascular access site disinfected with Alcohol(group1) and in group 2, Alcohol and povidone iodine 10% was used to separate were disinfected. Then the patient in a month of inflammation and infection of the vascular access will be monitor. Exclusion criteria: inflammation or fistula failure during the study for any reason other than infection. Sample size determination: Through the pilot study. Date: 02.10.2014 till 02.11.2014 Outcome: Washing with both solution affected on reduce the inflammation and infection of the patient.

the efficacy of Alcohol after Betadine and combination of alcohol and Betadine on inflammation and infection related to Vascular access hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* absence of inflammatory vascular access site
* three dialysis sessions per week

Exclusion Criteria:

* patient dies
* patient withdrew from the partnership

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
effected of betadin and alcohol on inflammation and infection of the patient | up to one month

CONTACTS AND LOCATIONS:
Overall Officials: mohmmad rajabpoor, student, Principal Investigator — Msc Student, Faculty of Nursing and Midwifery
Locations (1):
- Ali Bazzi, Mashhad, Iran

REFERENCES:
- [Background] Branas P, Morales E, Rios F, Sanz F, Gutierrez E, Quintanilla N, Orellana MA, Sanchez M, Rodriguez-Aranda A, Chaves F. Usefulness of endoluminal catheter colonization surveillance cultures to reduce catheter-related bloodstream infections in hemodialysis. Am J Infect Control. 2014 Nov;42(11):1182-7. doi: 10.1016/j.ajic.2014.07.022. Epub 2014 Sep 22. PMID 25248485
- See also: that is a article from pubmed — http://ncbi.nlm.nih.gov/pubmed/?term=hemodialysis+and+infection